CLINICAL TRIAL: NCT01105442
Title: Local Anaesthesia Used During Fast-track Colonic Surgery: Evaluation of Bupivacaine and Levobupivacaine in Practice
Status: Completed | Type: Observational
Sponsor: Martini Hospital Groningen (Other)
Responsible Party: Marinus van Hulst, Martini Hospital
Other Study IDs: METC2010-18
Record Dates: First submitted 2010-04-15; First posted 2010-04-16 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2010-03

CONDITIONS: Colonic Diseases; Post-operative Pain; Local Anesthesia
Keywords: Post-operative pain treatment; Fast-track colonic surgery patients; Surgery
MeSH Terms: conditions — Colonic Diseases; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Bupivacaine: Patients who received bupivacaine + sufentanil
- Levobupivacaine: Patients who received levobupivacaine and morphine on demand

SUMMARY:
The standard treatment for post operative pain is now bupivacaine + sufentanil. The use of this combination during fast-track colonic surgery leads frequently to post-operative nausea and vomiting and limited mobilisation possibilities. Therefore the department anaesthesiology wants to evaluate the use of a different local anaesthetic: levobupivacaine combined with morphine on demand. The expectation is that the use of levobupivacaine leads to less side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo fast-track colonic surgery and with post operative epidural pain treatment

Exclusion Criteria:

* Patients who are admitted to an other ward
* Patients with a spinal catheter

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Martini Hospital Groningen
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marinus van Hulst, Dr., Study Chair — Martini Hospital
Locations (1):
- Martini Hospital ward 4b, Groningen, Provincie Groningen, Netherlands